CLINICAL TRIAL: NCT02685514
Title: A Prospective Evaluation of High Intensity Focused Ultrasound (HIFU) in the Treatment of Relapsed Graves' Disease
Brief Title: A Evaluation of High Intensity Focused Ultrasound (HIFU) in the Treatment of Relapsed Graves' Disease
Acronym: HIFURGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Lang Hung Hin, Brian, Clinical Associate Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW16-015
Record Dates: First submitted 2016-02-14; First posted 2016-02-18 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Rrelapsed Graves' Disease
Keywords: HIFU; Graves' disease; treatment
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIFU Graves (Experimental): Applying the High intensity Focused Ultrasound treatment to the relapsed Graves' disease Patients.
  Interventions: Device: HIFU Graves

INTERVENTIONS:
Device: HIFU Graves — The HIFU treatment technique will be applied to the recruited participants

SUMMARY:
To evaluate the short-term efficiency and safety of HIFU treatment in the relapsed Graves' disease.

DETAILED DESCRIPTION:
Grave's disease is the most common cause of hyperthyroidism and affects approximately 2% of women and 0.2% of men in the population. The use of antithyroid drugs (ATD) has been the first-line of treatment for Graves' disease in many centers for decades, and its use has been increasing worldwide. One reason for this is that it may induce remission, whereas radioiodine (RAI) and surgery often lead to hypothyroidism and other complications in addition to hospitalization and radiation exposure. However, ATD use is also associated with increasing risk of some adverse minor effects such as skin rash, gastric intolerance, and arthralgia in 5% of patients. Furthermore, major adverse events, such as agranulocytosis and hepatotoxicity may be life-threatening but are rare (<0.5% of cases). These usually occur during the first three to six months of treatment, and tend to be associated with high ATD doses. Therefore, the recommended duration of ATD treatment is generally not longer than 12-24 months. However, despite adequate medical treatment, up to 50-70% of patients with Graves' disease would relapse or recur and therefore, a more definitive approach using RAI treatment or thyroid surgery is eventually needed for the resolution of hyperthyroidism. Although RAI is considered safe and easy to manage, particularly in patients without Grave's ophthalmopathy (GO), subclinical and overt hypothyroidism may occur months or even years after the administration of RAI. Hence, long-term follow-up of thyroid function and GO as well as management of thyroxine replacement is necessary. Similarly, although surgery is the main therapeutic strategy, it carries a 2%-10% risk of complications such as hypocalcemia, transient or permanent recurrent laryngeal nerve palsy, bleeding, or postoperative infection. In view of these, various nonsurgical, minimally invasive treatment alternatives have been developed at specialized treatment centers.

High-intensity focused ultrasound (HIFU) is a noninvasive procedure that involves application of a focused high-energy ultrasound beam for thermal tissue ablation inside the targeted zone, with minimal effect on the surrounding tissue. This method has been applied for treatment of a variety of medical conditions such as uterine fibroids and prostate, breast, pancreatic, and liver tumors. A favorable outcome also has been observed in patients with primary or secondary hyperparathyroidism. HIFU has also been proposed for thyroid nodule ablation . In a human feasibility study, 25 patients were treated 2 weeks before a scheduled thyroidectomy. Pathologic analysis demonstrated targeted tissue destruction of 2%-80% without any damage to neighboring structures. To the investigators knowledge, studies of follow-up after HIFU ablation of Graves' disease have not been published, except for one report where two patients received a combination of microwave ablation and RAI. Thus, the purpose of this prospective study is to assess the short-term efficacy and safety of US-guided HIFU ablation for the treatment of relapsed Graves' disease.

ELIGIBILITY:
Inclusion Criteria:

* age older than 18 years;
* relapsed Graves' disease despite an adequate ATD treatment for 18 months or more;
* HIFU accessibility of the targeted area (distance between the skin and the anterior surface of the nodule less than 10 mm; with no interference of the collarbone with HIFU unit movements);
* normal thyrotropin concentration before procedure;
* on at least 2-week of β-blockade prior to HIFU; and
* absence of vocal cord immobility at laryngoscopy.

Exclusion Criteria:

* patients who prefer or indicated for surgery;
* head and/or neck disease preventing hyperextension of the neck;
* history of thyroid cancer or other malignant tumors in the neck region;
* history of neck irradiation;
* severe Grave's ophthalmopathy (GO);
* large compressive goiter;
* pregnancy or lactation; and
* any contraindication related to intravenous moderate sedation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Remission rate of Graves' disease after one successful course of HIFU | 6 months
  To evaluate the remission rate of relapsed Graves' disease after 6 months of HIFU treatment

SECONDARY OUTCOMES:
The pain assessment (scoring 1-10) after treatment | 6 months
  Patient pain score immediately after HIFU treatment.
Incidence of local or general adverse events | 6 months
  The incidence rate of local or general adverse events after completion of HIFU treatment session.

CONTACTS AND LOCATIONS:
Overall Officials: Hung Hin, Brian Lang, MBBS(Hons), Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cooper DS. Antithyroid drugs. N Engl J Med. 2005 Mar 3;352(9):905-17. doi: 10.1056/NEJMra042972. No abstract available. PMID 15745981
- [Background] Watanabe N, Narimatsu H, Noh JY, Yamaguchi T, Kobayashi K, Kami M, Kunii Y, Mukasa K, Ito K, Ito K. Antithyroid drug-induced hematopoietic damage: a retrospective cohort study of agranulocytosis and pancytopenia involving 50,385 patients with Graves' disease. J Clin Endocrinol Metab. 2012 Jan;97(1):E49-53. doi: 10.1210/jc.2011-2221. Epub 2011 Nov 2. PMID 22049174
- [Background] Yip J, Lang BH, Lo CY. Changing trend in surgical indication and management for Graves' disease. Am J Surg. 2012 Feb;203(2):162-7. doi: 10.1016/j.amjsurg.2011.01.029. Epub 2011 Jun 17. PMID 21683939
- [Background] Zhou YF. High intensity focused ultrasound in clinical tumor ablation. World J Clin Oncol. 2011 Jan 10;2(1):8-27. doi: 10.5306/wjco.v2.i1.8. PMID 21603311
- [Background] Kovatcheva RD, Vlahov JD, Shinkov AD, Borissova AM, Hwang JH, Arnaud F, Hegedus L. High-intensity focused ultrasound to treat primary hyperparathyroidism: a feasibility study in four patients. AJR Am J Roentgenol. 2010 Oct;195(4):830-5. doi: 10.2214/AJR.09.3932. PMID 20858805
- [Background] Esnault O, Franc B, Chapelon JY. Localized ablation of thyroid tissue by high-intensity focused ultrasound: improvement of noninvasive tissue necrosis methods. Thyroid. 2009 Oct;19(10):1085-91. doi: 10.1089/thy.2009.0121. PMID 19803790
- [Background] Esnault O, Franc B, Menegaux F, Rouxel A, De Kerviler E, Bourrier P, Lacoste F, Chapelon JY, Leenhardt L. High-intensity focused ultrasound ablation of thyroid nodules: first human feasibility study. Thyroid. 2011 Sep;21(9):965-73. doi: 10.1089/thy.2011.0141. Epub 2011 Aug 11. PMID 21834683
- [Background] Esnault O, Franc B, Monteil JP, Chapelon JY. High-intensity focused ultrasound for localized thyroid-tissue ablation: preliminary experimental animal study. Thyroid. 2004 Dec;14(12):1072-6. doi: 10.1089/thy.2004.14.1072. PMID 15650361
- [Background] Korkusuz H, Happel C, Koch DA, Gruenwald F. Combination of Ultrasound-Guided Percutaneous Microwave Ablation and Radioiodine Therapy in Benign Thyroid Disease: A 3-Month Follow-Up Study. Rofo. 2016 Jan;188(1):60-8. doi: 10.1055/s-0041-106538. Epub 2015 Nov 13. PMID 26566268
- [Background] Huh JY, Baek JH, Choi H, Kim JK, Lee JH. Symptomatic benign thyroid nodules: efficacy of additional radiofrequency ablation treatment session--prospective randomized study. Radiology. 2012 Jun;263(3):909-16. doi: 10.1148/radiol.12111300. Epub 2012 Mar 21. PMID 22438360
- [Background] Kovatcheva RD, Vlahov JD, Stoinov JI, Kirilov GG, Krivoshiev SG, Arnaud F, Ortuno C, Drueke TB. High-intensity focussed ultrasound (HIFU) treatment in uraemic secondary hyperparathyroidism. Nephrol Dial Transplant. 2012 Jan;27(1):76-80. doi: 10.1093/ndt/gfr590. Epub 2011 Oct 19. PMID 22015443
- [Background] Kovatcheva R, Vlahov J, Stoinov J, Lacoste F, Ortuno C, Zaletel K. US-guided high-intensity focused ultrasound as a promising non-invasive method for treatment of primary hyperparathyroidism. Eur Radiol. 2014 Sep;24(9):2052-8. doi: 10.1007/s00330-014-3252-4. Epub 2014 Jun 4. PMID 24895038
- [Background] Esnault O, Rouxel A, Le Nestour E, Gheron G, Leenhardt L. Minimally invasive ablation of a toxic thyroid nodule by high-intensity focused ultrasound. AJNR Am J Neuroradiol. 2010 Nov;31(10):1967-8. doi: 10.3174/ajnr.A1979. Epub 2010 Jan 14. PMID 20075098